CLINICAL TRIAL: NCT02593032
Title: Study On The Effect of Combined Use of a Connected Pillbox, Pre-filled Medication Trays, Automated Text Message/Phone Call Reminds, On Medication Adherence in Patients With Type II Diabetes Mellitus, Hypertension or Hyperlipidemia
Brief Title: Effects of Use of a Connected Pillbox On Medication Adherence
Acronym: (TVHST2DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: TowerView Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 821737
Record Dates: First submitted 2015-10-19; First posted 2015-10-30 (Estimated); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus; Hypertension; Hyperlipidemia
Keywords: hemoglobin A1c protein, human > 7.5
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomized Treatment (Experimental): Patients in the treatment group will begin receiving their medications in pre-filled trays from Friendship Pharmacy. Patients will receive 5 trays on a monthly basis in order to accommodate a 30-day, insurance-reimbursed fill schedule.
  Interventions: Device: Pre-filled trays
- Control Arm (No Intervention): Patients in the control arm will receive usual care and can continue using their existing pharmacy.

INTERVENTIONS:
Device: Pre-filled trays — Randomized Control Trial Patients in the research treatment group receive pre-filled, 3x7 disposable trays that separate their medication by dose and time (e.g. morning, afternoon, evening). These pre-filled trays are inserted into a connected, weekly pillbox that detects when pills are removed from its wells.
  Arms: Randomized Treatment

SUMMARY:
Medication adherence is defined as the extent to which a patient takes his or her medication as prescribed by their healthcare provider. One third to one half of all patients in the United States do not take their medication as directed, resulting in nearly $100B in avoidable hospital costs per year. Recent efforts to improve medication adherence in patients with multiple comorbidities have turned to case management and disease management programs. Connected monitoring devices offer an alternative- or supplement- to frequent nurse visits and outreach. These devices enable frequent monitoring and intervention but can also generate large volumes of data that can be difficult for care teams to manage. The present study explores the use of one such device- a technology-enabled, connected pillbox. Given the continued emphasis on bending the cost curve in US healthcare, clinical validation of tools that may improve the management of costly chronic diseases, such as diabetes, is essential.

DETAILED DESCRIPTION:
Randomized Control Trial Patients in the research treatment group receive pre-filled, 3x7 disposable trays that separate their medication by dose and time (e.g. morning, afternoon, evening). These pre-filled trays are inserted into a connected, weekly pillbox that detects when pills are removed from its wells. Using this information, TowerView Health system is able to send automated text messages or phone reminders to patients to take forgotten or ignored medication doses. Medication adherence data from deployed pillboxes populates a software platform, which a research coordinator can access.

Patients who miss 3 consecutive doses or 5 doses out of 12 over a 4-day period trigger an alert for the study research coordinator who can contact the patient via phone call. The research coordinator follows a scripted motivational interview in his or her outreach to determine the etiology of non-adherence. Patients reporting worrisome symptoms will be instructed to contact their provider directly and/or go to the emergency room for immediate attention. The investigator acknowledges that the current study actually involves multiple interventions: 1. The pre-filled medication trays are provided by a pharmacist, which overcomes medication access issues as well as the inconvenience of manually organizing medications. 2. The electronic pillbox, which monitors adherence that triggers text message or phone reminders in instances where patients forget or ignore medication doses 3. Research coordinator alerts, which trigger outreach events that employ a motivational interview in order to improve patient adherence.

ELIGIBILITY:
Inclusion Criteria:• Insurance and pharmacy coverage with Independence Blue Cross (IBC); 18 years or older; Current diagnosis of Type II Diabetes Mellitus, Hypertension or Hyperlipidemia and taking 5 or more medications; Less than 80% medication adherence; Able to communicate in English; Willing to give informed consent, receive recruitment (invitation)letter from IBC

Exclusion Criteria: Known alcohol or illicit drug abuse; Significant cognitive impairment at baseline as defined by the Animal Naming Screening Tool; Residence in a care facility that provides medication on schedule; Unwilling to use TowerView Health's connected pillbox and accompanying medication trays; Any active medical or psychiatric diagnosis that, based on the clinical assessment of the research team, would prevent the study participant from completing the trial such as: markedly shortened life expectancy (e.g. diagnosis of metastatic cancer, end stage renal disease on dialysis, New York Heart Association (NYHA) Class III or IV heart failure, active psychosis or suicidal ideation, etc.) or dexterity/motor impairments (e.g. severe arthritis, neuromuscular disorders, etc); and Lack a mobile or land line phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2017-04 (Actual); Study Completion 2017-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nalaka S Gooneratne, MD, Principal Investigator — University of Pennsylvannia
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Randomized Treatment | Control Arm
Started | 17 | 33
Completed | 17 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Treatment | Control Arm | Total
Number analyzed (Participants) | 17 | 33 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (3.2) | 65 (3.4) | 64 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 25 | 36
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 24 | 35
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Self-reported adherence status to all medications [Number; unit: Number with self-reported low adherence] — Study participants were asked a single question that assessed their baseline self-reported adherence to any medications, with a 1 to 8 range of responses (Likert-type scale, 1=poor adherence and 8=high adherence), with a 6 or higher used to indicate "high adherence". This was assessed prior to beginning the study (i.e., a pre-treatment baseline assessment).
  Number with self-reported low adherence | 15 | 31 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Adherence at Month 6
Description: The primary outcome of interest in the present study is improvement in adherence. We will determine if a multi-modal intervention focused on improving medication adherence among adults who were previously non-adherent results in improved medication adherence over a 6-month interval averaged across months 1 to 6. This will be reported as the percent persistent on therapy at 6 months across the three conditions (diabetes, HTN, hyperlipidemia)
Time Frame: 6-month interval
Measure: Number; unit: percent persistent on therapy
Arm/Group | Randomized Treatment | Control Arm
Number analyzed (Participants) | 17 | 33
percent persistent on therapy | 91 | 40
Statistical Analysis 1: Comparison: Randomized Treatment vs Control Arm; Test type: Superiority; p < 0.05, t-test, 2 sided — This is the calculated p-value, not a threshold; Mean Difference (Net) = 12

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Randomized Treatment | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/33
Other Adverse Events (participants affected / at risk) | 0/17 | 0/33

LIMITATIONS AND CAVEATS:
Early termination due to funding constraints, leading to a smaller sample size than originally proposed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT02593032/Prot_SAP_000.pdf